CLINICAL TRIAL: NCT00141245
Title: Pregabalin Open-Label, Multicenter Add-On Trial Following a 4-Day Double-Blind Transition Period to Determine Long-Term Safety and Efficacy in Patients With Partial Seizures.
Brief Title: To Evaluate Long-Term Safety and Efficacy of Pregabalin in Patients With Partial Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-012
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: Seizure Disorder, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate long-term safety and efficacy of pregabalin in patients with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for preceding double-blind study
* Have received double-blind study medication and wish to receive open-label pregabalin.

Exclusion Criteria:

* Cannot have absence seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325
Dates: Start 1998-10; Study Completion 2005-11

PRIMARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- Australia (6):
  - Pfizer Investigational Site, Deakin, Australian Capital Territory
  - Pfizer Investigational Site, Chatswood, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Woodville
- Austria (2):
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Innsbruck
- Pfizer Investigational Site, Duffel, Belgium
- Finland (2):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Turku
- France (6):
  - Pfizer Investigational Site, Lyon, Cedex
  - Pfizer Investigational Site, Paris, Cedex
  - Pfizer Investigational Site, Tours, Cedex
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Roubaix
- Germany (8):
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Mönchengladbach
  - Pfizer Investigational Site, Munich
  - Pfizer Investigational Site, Münster
- Italy (4):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
- Netherlands (2):
  - Pfizer Investigational Site, Heemstede
  - Pfizer Investigational Site, Heeze
- South Africa (2):
  - Pfizer Investigational Site, Parow, Cape Town
  - Pfizer Investigational Site, Durban
- Spain (4):
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Barcelona
- Pfizer Investigational Site, Gothenburg, Sweden
- Switzerland (2):
  - Pfizer Investigational Site, Lavigny, LE
  - Pfizer Investigational Site, Tschugg
- United Kingdom (6):
  - Pfizer Investigational Site, Bimingham
  - Pfizer Investigational Site, Bucks
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, York